CLINICAL TRIAL: NCT04908917
Title: Reducing AIR Pollution Exposure to Lower Blood PRESSURE
Brief Title: Reducing Air Pollution to Lower Blood Pressure
Acronym: AIR PRESSURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Youcheng Liu, Associate Professor, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-21-05-3595
Record Dates: First submitted 2021-05-22; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Mild Hypertension; Air Pollution Exposure

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, double-blind, sham-controlled parallel limb clinical trial. Two-hundred participants will be recruited and randomly allocated into the intervention group (N=100) to use a PAC with a HEPA filter in the bedroom and the control group (N=100) with a sham PAC (no HEPA filter inside the container).
Who Masked: Participant, Investigator
Masking Description: Once a participant is recruited, an identification number in a sequence number (001, 002, 003, etc.) will be assigned to him or her. A simple randomization will be performed by the unblind study Biostatistician with random block sizes of 4 and 6 to allocate recruited participants into the intervention group (N=100, 50% allocation rate, PAC use with HEPA filter) and control group (N=100, allocation rate 50%, PAC use without HEPA filter).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAC with HEPA (Experimental): Intervention group (N=100) to use a portable air cleaner (with a HEPA filter in PAC)
  Interventions: Device: Portable Air Cleaner with a HEPA Filter
- PAC without HEPA (Sham Comparator): control group (N=100) with a sham portable air cleaner (no HEPA filter in PAC)
  Interventions: Device: Portable Air Cleaner without a HEPA Filter

INTERVENTIONS:
Device: Portable Air Cleaner with a HEPA Filter — A novel intervention using a portable air cleaner with HEPA filter to treat mildly high BP to potentially reduce the cardiovascular effects of PM2.5. Leave the PAC running with the HEPA filter installed on the highest setting during sleeping periods in the room in which the participant sleeps.
  Arms: PAC with HEPA
Device: Portable Air Cleaner without a HEPA Filter — Leave the PAC running without a HEPA filter installed on the highest setting during sleeping periods in the room in which the participant sleeps.
  Other Names: Control
  Arms: PAC without HEPA

SUMMARY:
Fine particulate matter <2.5 μm (PM2.5) air pollution is the fifth leading risk factor for global mortality. Mitigating the clinically significant blood pressure (BP) elevation from air pollution by reducing PM2.5 exposure will likely contribute to the reduction in cardiovascular disease-related mortality. Twin epidemics of air pollution and high BP converge in underserved urban communities (i.e., Detroit) and warrant immediate attention. Prior studies with short duration (a few days) showed indoor portable air cleaners (PACs) are a novel approach to reduce the health burden of both high BP and PM2.5. Trials over several weeks employing remote technologies with a large sample size of patients residing in their own homes in vulnerable urban communities are needed to demonstrate if the BP-reduction from PAC usage is sustainable in real-world settings. The investigators' specific aims are to 1) determine if compared to sham, active PAC use during 3 weeks can provide sustained reductions in home BP levels by reducing personal-level PM2.5 air pollution exposures in patients with mild high BP residing in vulnerable disadvantaged communities across Detroit and 2) explore clinical markers (e.g., age, sex, body mass index) that predict BP-responses to PAC intervention to better target at-risk populations in larger-scale trials and future real-world clinical settings. A randomized, double-blind, sham-controlled parallel limb trial of overnight bedroom PAC use versus sham with 200 Detroit community individuals with mild high BP will be conducted. Continuous bedroom PM2.5 levels and home BP will be measured throughout 28 days. PAC will be used in the bedroom before bedtime on the 7th day continuously for 21 days. The reduction of systolic BP (SBP) will be calculated for both the intervention and control groups and the significance will be compared using mixed-effects modeling with repeated measurements of SBP as the dependent variable and group (active vs sham PAC use) as the independent variable with a fixed-effect. Linear multiple regression modeling with SBP as the dependent variable and participant-level characteristics including body mass index, waist circumference, race, ethnicity, or sex as predictors will be explored. This study is expected to demonstrate a significant sustainable reduction in home SBP for active PAC vs sham use in this population with mildly high BP.

DETAILED DESCRIPTION:
1. Air pollution caused by fine particulate matter with aerodynamic diameter <2.5 μm (PM2.5) is the fifth leading risk factor for global mortality,1,2 predominantly due to cardiovascular disease (CVD).3-5 While several mechanisms are responsible,4,6 PM2.5-induced elevations in blood pressure (BP) was identified as a key pathway.7-10 Short term (hours-days) PM2.5 exposures increase systolic BP (SBP) by 2-10 mmHg in a dose-dependent manner while longer term exposures (months-to-years) promote the onset of hypertension (HTN).7,11,12 Relevant mechanisms include systemic inflammation, autonomic and vascular dysfunction, and activation of the renin-angiotensinaldosterone system (RAAS).4,5,7 Recent estimates of annual PM2.5 mortality are 8.9 million globally, due in part to PM2.5-mediated HTN.1,13 Exposure to current levels of ambient PM2.5 in the U.S. is associated with elevated BP, increased CVD risk and an estimated 213,000 deaths annually.1 Given the billions of people impacted, PM2.5 is an independent (modifiable) HTN risk factor of global public health importance. Therefore, mitigating the clinically significant BP elevation from air pollution by reducing PM2.5 exposure will likely contribute to the reduction in CVD-related mortality.
2. HTN is the leading risk factor for global morbidity and mortality and a major cause of health disparities. Nearly 50% of US adults meet criteria (≥130/80 mm Hg) for HTN.14 Serious disparities persist such that underserved communities, including Detroit, have the highest prevalence of HTN and the poorest treatment success. Mounting evidence indicates that PM2.5 contributes to this epidemic of HTN,7-11 and that individuals in disadvantaged urban environments (e.g., Detroit) face higher concentrations of air pollutants.15-17 Low socioeconomic status communities are especially "vulnerable" (i.e., highly exposed) and "susceptible" (i.e., higher risk for adverse health effects) to air pollution.15,17,18 In Detroit, CV mortality has been shown to be jointly impacted by high PM2.5 levels and vulnerability to exposures in communities of color and lower socioeconomic status. The investigators' studies have shown that air pollutants in the city of Detroit are responsible for increasing BP. Hence, addressing the co-epidemics of PM2.5 exposure and cardiometabolic illnesses is not only an issue of public health importance but also of environmental justice for urban settings such as Detroit. Thus, the twin epidemics of air pollution and HTN converge in underserved urban communities (i.e., Detroit) and warrant immediate attention. The novel recruitment strategy using the Wayne State University (WSU) mobile health units (MHUs) directly reaches out to disadvantaged communities across Detroit so those disproportionally affected by PM2.5 and high BP can be enrolled.
3. Indoor portable air cleaners (PACs) are a novel approach to reduce the health burden of both HTN and PM2.5. In a meta-analysis of 10 PAC trials (n=604), it was shown that a ≈30-60% reduction in PM2.5 lowered SBP by ≈4 mm Hg over ≈13 days.19 In the investigators' trial of 40 nonsmokers living in urban senior housing,20 PACs lowered personal PM2.5 by ≈40% and morning SBP by 3.2 mmHg over 3 days, with greater reductions (≈8 mm Hg) in obese individuals. Emerging evidence shows that obesity and underlying cardiometabolic abnormalities play a mechanistic role in PM2.5-induced BP elevations and may underlie their susceptibility to PM2.5 and heightened BP-lowering responsiveness to PACs. This supports that populations commonly suffering from obesity, including African American hypertensives, may gain especially potent benefits from PACs. Trials over several weeks employing remote technologies with a large sample size of patients residing in their own homes in vulnerable urban communities are needed to demonstrate if the BP-reduction from PAC usage is sustainable in real-world settings. These are the features and innovations of the current study.

Prior studies in air pollution exposure intervention all have used physical contact methods with participants to assess exposure and measure BP. However, such direct contact and home visit methods to collect data during this COVID-19 pandemic becomes a challenge and unsafe for both investigators and study participants. Additionally, it costs more manpower and resources. Modern monitoring techniques, equipment and communication technologies provide data collection using a "low touch" method of remote monitoring of PM-reduction and home BP (HBP) lowering which is important in COVID era as well as to reduce patient burden and reduce patient follow-up. This will lend itself to be potentially greatly upscaled if patients can do all endpoints via remote technology. This study will be the first to test this technology as it applies to epidemiologic studies. This has never been tested before.

Additionally, studies in past used mixed populations with different BP levels and disease status. It is not known if reducing BP by reducing PM2.5 exposure using PACs also will work on people with mild HTN. In this study, the investigators' will focus specifically on people with mild HTN -the patients who actually need BP-lowering intervention for early treatment. This has not been looked at in this mild HTN population.

This study will serve as a pivotal trial to demonstrate that PACs are: 1) an effective method to lower PM2.5 exposure and SBP; and 2) a novel intervention to treat mild high BP and potentially reduce the cardiovascular effects of PM2.5. 3) The investigators' aim to show that novel low-touch remote methods are acceptable and reliable for assessing the benefits of air pollution interventions and that they could be expanded to thousand participants and benefit large number of vulnerable community members.

The current study has several key innovations and contributions. This will be the first PAC trial to: 1) Persist longer than a few days in intervention duration, allowing us to determine if BP reduction with PAC use is sustainable over a clinically relevant duration of 21 days of active use. 2) This trial is ≈ 5-fold larger than the earlier trial in Detroit in order to provide the most definitive evidence ("pivotal trial") and allow for testing of effect modifiers (e.g., obesity) in medium-risk populations with mild high BP most likely to benefit from a novel BP lowering intervention. 3) Leverage existing WSU MHUs to address environmental inequities for urban patients with high BP. 4) Employ mobile technologies and remote monitoring to capture home BP and PM2.5 levels via "low-touch" methods in a real-world community setting in patients vulnerable to the health effects of high BP and PM2.5 exposures.

The investigators hypothesize that 1) PAC use will reduce indoor exposure to PM2.5 which will subsequently reduce SBP. 2) This reduction in home BP will be sustainable over several weeks in people with mildly high BP. 3) The study can be conducted via "low touch" remote technology (using home BP and PM monitors). 4) This remote technology will be employable and acceptable to vulnerable members of disadvantaged communities across Detroit.

Primary Aim: To determine if compared to sham, active PAC use during clinically relevant periods can provide sustained reductions in HBP levels (over 21 days) by reducing personal-level fine particulate matter (PM2.5) air pollution exposures in patients with mildly high BP residing in vulnerable disadvantaged communities across Detroit.

Secondary Aim: To explore clinical biomarkers (age, sex, body mass index) that predict the BP-lowering response to PAC intervention to target at-risk populations in larger-scale interventions and future real-world clinical settings and future real-world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported nonsmokers (for at least last year)
* Has own smartphone
* Systolic BP (SBP) at 120-145 mmHg
* Diastolic blood pressure (DBP) <95 mmHg
* Has history of hypertension with ≤ 3 medications and stable without change in past 3 months
* If medications are used, there should be no change in dosage during the 28-day study period.

Exclusion Criteria:

* Living with an active smoker who smokes indoors
* Left upper arm circumference >17 inches (measured by tape measure upon recruitment as needed as it makes the home BP device inaccurate)
* Pregnant
* Unable/unwilling to consent
* Established cardiovascular disease (CVD)
* Stage IV clinical kidney disease (CKD)
* Clear barrier to technology use (e.g., visual or hearing impairment)
* Lung disease requiring oxygen
* Cancer receiving treatment
* Diabetes
* COVID-19 infections
* Any condition where the investigators believe the risk of a mildly high BP above 130/80 mmHg may pose risk to the patient during the 28-day period of the study including but not limited to aortic aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure change measured by blood pressure meter | 28 days (Day 1 to Day 28 of the 4-week study).
  Home systolic and diastolic blood pressures will be measured using a self-administered blood pressure meter before (7 days) and during (21 days) the use of a portable air cleaner and compared between before and during use to see if blood pressures will be reduced during the air cleaner use phase, and between the intervention and control groups to see if there is a difference in blood pressure reduction between the two groups.

SECONDARY OUTCOMES:
Demographaic characteristics measured by a questionnaire | One-time measurement at baseline (Day 1 to Day 7)
  Demographic characteristics such as age, sex, race/ethnicity and education will be measured using a questionnaire. All these variables will be assessed to see if they predict the blood pressure reduction (Primary Outcome).
Body mass index (BMI) | One-time measurement (Day 1 to Day 7)
  Height and weight will be measured using a scale and tape measured and combined to report BMI in kg/m^2. BMI will be assessed to see if it predicts the blood pressure reduction (Primary Outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Youcheng Liu, MD, ScD, MS, MPH, Principal Investigator — Wayne State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burnett R, Chen H, Szyszkowicz M, Fann N, Hubbell B, Pope CA 3rd, Apte JS, Brauer M, Cohen A, Weichenthal S, Coggins J, Di Q, Brunekreef B, Frostad J, Lim SS, Kan H, Walker KD, Thurston GD, Hayes RB, Lim CC, Turner MC, Jerrett M, Krewski D, Gapstur SM, Diver WR, Ostro B, Goldberg D, Crouse DL, Martin RV, Peters P, Pinault L, Tjepkema M, van Donkelaar A, Villeneuve PJ, Miller AB, Yin P, Zhou M, Wang L, Janssen NAH, Marra M, Atkinson RW, Tsang H, Quoc Thach T, Cannon JB, Allen RT, Hart JE, Laden F, Cesaroni G, Forastiere F, Weinmayr G, Jaensch A, Nagel G, Concin H, Spadaro JV. Global estimates of mortality associated with long-term exposure to outdoor fine particulate matter. Proc Natl Acad Sci U S A. 2018 Sep 18;115(38):9592-9597. doi: 10.1073/pnas.1803222115. Epub 2018 Sep 4. PMID 30181279
- [Result] Cohen AJ, Brauer M, Burnett R, Anderson HR, Frostad J, Estep K, Balakrishnan K, Brunekreef B, Dandona L, Dandona R, Feigin V, Freedman G, Hubbell B, Jobling A, Kan H, Knibbs L, Liu Y, Martin R, Morawska L, Pope CA 3rd, Shin H, Straif K, Shaddick G, Thomas M, van Dingenen R, van Donkelaar A, Vos T, Murray CJL, Forouzanfar MH. Estimates and 25-year trends of the global burden of disease attributable to ambient air pollution: an analysis of data from the Global Burden of Diseases Study 2015. Lancet. 2017 May 13;389(10082):1907-1918. doi: 10.1016/S0140-6736(17)30505-6. Epub 2017 Apr 10. PMID 28408086
- [Result] Newby DE, Mannucci PM, Tell GS, Baccarelli AA, Brook RD, Donaldson K, Forastiere F, Franchini M, Franco OH, Graham I, Hoek G, Hoffmann B, Hoylaerts MF, Kunzli N, Mills N, Pekkanen J, Peters A, Piepoli MF, Rajagopalan S, Storey RF; ESC Working Group on Thrombosis, European Association for Cardiovascular Prevention and Rehabilitation; ESC Heart Failure Association. Expert position paper on air pollution and cardiovascular disease. Eur Heart J. 2015 Jan 7;36(2):83-93b. doi: 10.1093/eurheartj/ehu458. Epub 2014 Dec 9. No abstract available. PMID 25492627
- [Result] Rajagopalan S, Al-Kindi SG, Brook RD. Air Pollution and Cardiovascular Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2018 Oct 23;72(17):2054-2070. doi: 10.1016/j.jacc.2018.07.099. PMID 30336830
- [Result] Brook RD, Newby DE, Rajagopalan S. Air Pollution and Cardiometabolic Disease: An Update and Call for Clinical Trials. Am J Hypertens. 2017 Dec 8;31(1):1-10. doi: 10.1093/ajh/hpx109. PMID 28655143
- [Result] Bevan GH, Al-Kindi SG, Brook RD, Munzel T, Rajagopalan S. Ambient Air Pollution and Atherosclerosis: Insights Into Dose, Time, and Mechanisms. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):628-637. doi: 10.1161/ATVBAHA.120.315219. Epub 2020 Dec 17. PMID 33327745
- [Result] Giorgini P, Di Giosia P, Grassi D, Rubenfire M, Brook RD, Ferri C. Air Pollution Exposure and Blood Pressure: An Updated Review of the Literature. Curr Pharm Des. 2016;22(1):28-51. doi: 10.2174/1381612822666151109111712. PMID 26548310
- [Result] Cai Y, Zhang B, Ke W, Feng B, Lin H, Xiao J, Zeng W, Li X, Tao J, Yang Z, Ma W, Liu T. Associations of Short-Term and Long-Term Exposure to Ambient Air Pollutants With Hypertension: A Systematic Review and Meta-Analysis. Hypertension. 2016 Jul;68(1):62-70. doi: 10.1161/HYPERTENSIONAHA.116.07218. Epub 2016 May 31. PMID 27245182
- [Result] Liang R, Zhang B, Zhao X, Ruan Y, Lian H, Fan Z. Effect of exposure to PM2.5 on blood pressure: a systematic review and meta-analysis. J Hypertens. 2014 Nov;32(11):2130-40; discussion 2141. doi: 10.1097/HJH.0000000000000342. PMID 25250520
- [Result] Yang BY, Qian Z, Howard SW, Vaughn MG, Fan SJ, Liu KK, Dong GH. Global association between ambient air pollution and blood pressure: A systematic review and meta-analysis. Environ Pollut. 2018 Apr;235:576-588. doi: 10.1016/j.envpol.2018.01.001. Epub 2018 Jan 11. PMID 29331891
- [Result] Dvonch JT, Kannan S, Schulz AJ, Keeler GJ, Mentz G, House J, Benjamin A, Max P, Bard RL, Brook RD. Acute effects of ambient particulate matter on blood pressure: differential effects across urban communities. Hypertension. 2009 May;53(5):853-9. doi: 10.1161/HYPERTENSIONAHA.108.123877. Epub 2009 Mar 9. PMID 19273743
- [Result] Brook RD, Bard RL, Burnett RT, Shin HH, Vette A, Croghan C, Phillips M, Rodes C, Thornburg J, Williams R. Differences in blood pressure and vascular responses associated with ambient fine particulate matter exposures measured at the personal versus community level. Occup Environ Med. 2011 Mar;68(3):224-30. doi: 10.1136/oem.2009.053991. Epub 2010 Oct 8. PMID 20935292
- [Result] Lelieveld J, Evans JS, Fnais M, Giannadaki D, Pozzer A. The contribution of outdoor air pollution sources to premature mortality on a global scale. Nature. 2015 Sep 17;525(7569):367-71. doi: 10.1038/nature15371. PMID 26381985
- [Result] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Result] Hajat A, Allison M, Diez-Roux AV, Jenny NS, Jorgensen NW, Szpiro AA, Vedal S, Kaufman JD. Long-term exposure to air pollution and markers of inflammation, coagulation, and endothelial activation: a repeat-measures analysis in the Multi-Ethnic Study of Atherosclerosis (MESA). Epidemiology. 2015 May;26(3):310-20. doi: 10.1097/EDE.0000000000000267. PMID 25710246
- [Result] Di Q, Wang Y, Zanobetti A, Wang Y, Koutrakis P, Choirat C, Dominici F, Schwartz JD. Air Pollution and Mortality in the Medicare Population. N Engl J Med. 2017 Jun 29;376(26):2513-2522. doi: 10.1056/NEJMoa1702747. PMID 28657878
- [Result] Bowe B, Xie Y, Yan Y, Al-Aly Z. Burden of Cause-Specific Mortality Associated With PM2.5 Air Pollution in the United States. JAMA Netw Open. 2019 Nov 1;2(11):e1915834. doi: 10.1001/jamanetworkopen.2019.15834. PMID 31747037
- [Result] Martenies SE, Milando CW, Williams GO, Batterman SA. Disease and Health Inequalities Attributable to Air Pollutant Exposure in Detroit, Michigan. Int J Environ Res Public Health. 2017 Oct 19;14(10):1243. doi: 10.3390/ijerph14101243. PMID 29048385
- [Result] Walzer D, Gordon T, Thorpe L, Thurston G, Xia Y, Zhong H, Roberts TR, Hochman JS, Newman JD. Effects of Home Particulate Air Filtration on Blood Pressure: A Systematic Review. Hypertension. 2020 Jul;76(1):44-50. doi: 10.1161/HYPERTENSIONAHA.119.14456. Epub 2020 Jun 1. PMID 32475316
- [Result] Morishita M, Adar SD, D'Souza J, Ziemba RA, Bard RL, Spino C, Brook RD. Effect of Portable Air Filtration Systems on Personal Exposure to Fine Particulate Matter and Blood Pressure Among Residents in a Low-Income Senior Facility: A Randomized Clinical Trial. JAMA Intern Med. 2018 Oct 1;178(10):1350-1357. doi: 10.1001/jamainternmed.2018.3308. PMID 30208394